CLINICAL TRIAL: NCT00599547
Title: Allogeneic Stem Cell Transplantation After Dose-reduced Intensity Conditioning Regimen for Patients With Myelofibrosis With Myeloid Metaplasia (MMM): A Phase II-study
Brief Title: Allogeneic Stem Cell Transplantation (SCT) After Dose-reduced Conditioning for Myelofibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBMT AlloRIC-MMM
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Myelofibrosis
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic Stem Cell Transplantation (Experimental): Allogeneic Stem Cell Transplantation after dose-reduced Conditioning for Myelofibrosis Patients
  Interventions: Procedure: Allogeneic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Allogeneic Stem Cell Transplantation — Allogeneic Stem Cell Transplantation after dose-reduced Conditioning for Myelofibrosis Patients

SUMMARY:
The purpose of this study is to determine whether a reduced intensity conditioning regimen followed by allogeneic stem cell transplantation is a feasible and effective treatment for patients with primary myelofibrosis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a reduced intensity conditioning regimen followed by allogeneic stem cell transplantation from related or unrelated donors is a feasible and effective treatment for patients with primary myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Disease: Histologically proven Myelofibrosis with myeloid metaplasia/MMM defined as per the Italian Consensus Conference on MMM diagnosis with either primary MMM or secondary to Polycythaemia vera or essential thrombocythaemia with

  * "intermediate risk" or "high risk" score according to the Lille Scoring System
  * OR "low risk" score according to the Lille Scoring System with constitutional symptoms (fever, night sweat, weight loss > 5% of body weight)
  * OR "high risk" score according to the Cervantes score
* Age:

  * Patients between 50 and 70 years of age and no limited life expectancy for other reasons than MMM
  * Patients under 50 years of age who are not eligible for a standard myeloablative conditioning, (e.g., because of prior autologous stem cell, history of severe infections like fungal infections, history of cardiac toxicity or other reasons according to the treating physician)
* HLA compatible or identical donor, related or unrelated (one mismatch allowed)
* Written informed consent of the patient

Exclusion Criteria:

* Positive search for bcr-abl on blood.
* Serious irreversible renal, hepatic, pulmonary or cardiac disease
* Central nervous involvement
* Positive serology for HIV
* Pregnant or lactating women
* Patients with a life-expectancy of less than six months because of another debilitating disease
* Serious psychiatric or psychological disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2002-11; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality by day +100 and by one year post-transplant, hematopoietic recovery by day +100 post-transplant, myeloid and T-cell chimerism by day +100 posttransplant, toxicity of the regimen acc. to Bearman scale | Follow-up until day +1095

SECONDARY OUTCOMES:
VOD-Staging and VOD-Grading acc. to the McDonald-scale, incidence of GvHD, overall survival post-transplant, disease-free survival post-transplant | Follow-up until day +1095

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Kroger N, Holler E, Kobbe G, Bornhauser M, Schwerdtfeger R, Baurmann H, Nagler A, Bethge W, Stelljes M, Uharek L, Wandt H, Burchert A, Corradini P, Schubert J, Kaufmann M, Dreger P, Wulf GG, Einsele H, Zabelina T, Kvasnicka HM, Thiele J, Brand R, Zander AR, Niederwieser D, de Witte TM. Allogeneic stem cell transplantation after reduced-intensity conditioning in patients with myelofibrosis: a prospective, multicenter study of the Chronic Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Blood. 2009 Dec 17;114(26):5264-70. doi: 10.1182/blood-2009-07-234880. Epub 2009 Oct 7. PMID 19812383